CLINICAL TRIAL: NCT04110132
Title: Postoperative Analgesia Using Ganglion Impar Block After Anal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16/70-8/2/2017
Record Dates: First submitted 2018-05-05; First posted 2019-10-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: After approval of local ethical committee and patient consent, this double blinded randomized study will be done on 60 patients undergoing hemorrhoidectomy surgery in Alexandria University hospital.
  After standard general anesthesia with Propofol 1-2mg/kg LMA for airway management and maintenance with Isoflurane 1%. The patient will be randomized into two groups.
  Bupivacaine group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Bupivacaine 0.5% 10ml.
  Saline group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Normal Saline 10ml
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant, care provider and outcomes assessors will not be aware of the used intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ganglion impar block with Bupivacaine. (Active Comparator): Bupivacaine group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Bupivacaine 0.5% 10ml.
  Patient will have hemorrhoidectomy.
  Interventions: Procedure: Ganglion impar block with Bupivacaine.
- Ganglion impar block with Saline (Placebo Comparator): Saline group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Normal Saline 10ml Patient will have hemorrhoidectomy.
  Interventions: Procedure: Ganglion impar block with normal saline

INTERVENTIONS:
Procedure: Ganglion impar block with Bupivacaine. — Bupivacaine group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Bupivacaine 0.5% 10ml.
  Postoperative VAS will be measured each 1 for the first 6 hours then at 9 and 12 hours postoperative.
  Arms: Ganglion impar block with Bupivacaine.
Procedure: Ganglion impar block with normal saline — Saline group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Normal Saline 10ml Postoperative VAS will be measured each 1 for the first 6 hours then at 9 and 12 hours postoperative.
  Arms: Ganglion impar block with Saline

SUMMARY:
The aim of this study is to evaluate the ganglion Impar block in the prevention of postoperative pain after anal surgery.

DETAILED DESCRIPTION:
Postoperative analgesia using ganglion Impar block after anal surgery

Introduction

Ganglion Impar block may be used for treatment of chronic perineal pain (1) Aim

The aim of this study is to evaluate the ganglion Impar block in the prevention of postoperative pain after anal surgery.

Patients and Methods

After approval of local ethical committee and patient consent, this double blinded randomized study will be done on 60 patients undergoing hemorrhoidectomy surgery in Alexandria University hospital.

After standard general anesthesia with Propofol 1-2mg/kg LMA for airway management and maintenance with Isoflurane 1%. The patient will be randomized into two groups.

Bupivacaine group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Bupivacaine 0.5% 10ml.

Saline group; Ganglion Impar will be blocked using G25 Quinqe spinal needle using Normal Saline 10ml Postoperative VAS will be measured each 1 for the first 6 hours then at 9 and 12 hours postoperative.

First request of pain medications will be measured.

Results Results will be collected in tables and graphs. Appropriate statistical analysis will be done.

Discussion Results of the study will be discussed compared to other studies.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hemorrhoidectomy surgery in Alexandria University hospital.

Exclusion Criteria:

* Coagulation effects
* Allergy to Bupivacaine
* Previous anal surgery
* Patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2028-07-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  VAS sore 0-10

SECONDARY OUTCOMES:
First request of pain medications will be measured. | 24 hours
  Time in hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardaillac C, Ploteau S, Labat JJ, Levesque A, Riant T. [Interest of infiltration of Impar node in rebel vulvodynia: About a series of 8 cases]. Prog Urol. 2016 Dec;26(17):1213-1221. doi: 10.1016/j.purol.2016.08.004. Epub 2016 Sep 7. French. PMID 27614384